CLINICAL TRIAL: NCT04902287
Title: From Science to Practice: An Evidence Based Engagement Intervention to Support Treatment Success for Youth's Problematic Sexual Behavior
Brief Title: PHF Problematic Sexual Behavior of Youth Family Engagement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ending due to PI leaving position at the University of Oklahoma.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20211217
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Trauma, Sexual
MeSH Terms: conditions — Sexual Trauma

STUDY DESIGN:
Intervention Model Description: The current clinical trial involves two conditions (N=20 each): engagement condition or referral as usual
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIES Engagement Strategies (Experimental): Participants in this arm will receive a 30-minute TIES engagement intervention during their referral phone call.
  Interventions: Behavioral: Training Intervention for the Engagement of Families (TIES)
- Referral as Usual (No Intervention): Participants in this arm will receive a standard call to schedule an intake appointment by an administrative assistant with no clinical training.

INTERVENTIONS:
Behavioral: Training Intervention for the Engagement of Families (TIES) — This intervention involves training service personnel in a method of communication that elicits a person's intrinsic motivation for change.
  Arms: TIES Engagement Strategies

SUMMARY:
Efficacious child mental health services are only helpful if families engage in services; however, as many as 75% of families in need never establish contact with a mental health professional and greater than half of families fail to attend their first appointment. Fortunately, interventions have been developed to increase the likelihood that families will participate in treatment. Despite the development of these interventions, no research to date has evaluated these strategies with a critically important population, youth with problematic sexual behaviors (PSB). PSBs in children are a substantial public health concern, as greater than one-third of child sexual abuse cases are committed by other youth. Evidence based practices (EBP's) that include direct engagement of caregivers in services for youth PSB have strong efficacy, with recidivism rates of two percent. Thus, a therapeutic response that successfully engages families is necessary to promote community safety. Research has indicated that engagement of families in PSB treatment has greater complications due to managing internal and external experiences of shame, stigma, and misperceptions of youth. Therefore, the present study seeks to determine the impact of a first contact intervention to assess if strategies aid in the engagement of families in treatment for youth PSB as compared to referral as usual. This will be accomplished by conducting a small-scale Randomized Control Trial. This project is the first step in an innovative line of research that will provide practical strategies for practitioners to utilize in order to successfully recruit, retain, and heal families of youth with PSB.

DETAILED DESCRIPTION:
Efficacious child mental health services are only helpful if families engage in services. However, as many as 75% of families in need never establish contact with a mental health professional and greater than half of families fail to attend their first scheduled visit. Fortunately, first contact interventions have reduced barriers and increased the likelihood that a family begin services following initial referral. Research has demonstrated the effectiveness of a phone intervention using 'Training Intervention for the Engagement of Families' (TIES) for engagement of families referred to outpatient behavioral health services due to childhood trauma and disruptive behavior disorders. However, engagement intervention strategies have not yet been applied to a critically important population, youth with problematic sexual behaviors (PSB), who face unique barriers to engagement in treatment. PSBs in children are a substantial public health concern, as greater than one-third of child sexual abuse cases have been found to be committed by other youth. Evidence based practices (EBP's) that include direct engagement of caregivers in services for children with PSB have strong efficacy, with recidivism rates of two percent. Thus, a therapeutic response is most logical to promote community safety and prevent future incidence of PSB. Despite the development of efficacious treatment, EBP's are not provided to most youth with PSB. Our research has indicated that engagement of families when a child has PSB has greater complications due to managing internal and external experiences of shame, stigma, and misperceptions surrounding the youth's behaviors, as well as navigation of a large number of systems (e.g., child welfare, juvenile justice, law enforcement). Given the potential negative impact of treatment attrition on overall community safety and child well-being, research efforts concentrated on identifying strategies that enhance service engagement for the treatment of youth with PSB are warranted. While TIES strategies have shown great promise in increasing family engagement, no research to date has examined the impact of purposeful, evidence-based engagement intervention on decreasing attrition amongst families of youth with PSB. A critical gap exists in the research literature, as families of youth with PSB face additional perceptual barriers to engaging in treatment such as a hesitancy to discuss stigmatizing behaviors due to feelings of responsibility and shame. Therefore, the present study seeks to determine the impact of this intervention to assess if these strategies successfully aid in both the successful engagement of families in treatment for youth PSB as compared to referral as usual. This will be accomplished by conducting a small-scale Randomized Control Trial (RCT). We will test the hypothesis that TIES engagement strategies will improve both initial and sustained engagement in EBP as compared to referral as usual amongst families of school aged children with PSB. The proposed study will accomplish this through the following specific aims:

Aim 1. To examine the efficacy of an evidence-based engagement intervention strategy for successfully engaging families of youth with PSB in treatment. Families' who are referred to the PSB-CBT treatment services will be randomly assigned to TIES strategies or referral as usual procedures to test the impact of an evidence-based engagement intervention on program attrition. Factors such as parenting stress, child emotional and behavioral health concerns, treatment satisfaction and alliance will be examined to understand their unique contribution to family attrition in treatment for this population.

Aim 2. In order to accomplish Aim 1, we will first systematically adapt the TIES intervention to meet the unique needs of families of youth with PSB to improve the ability of TIES to decrease overall attrition. Adaptations to TIES strategies will include supporting families to overcome barriers such as navigating community systems and addressing misperceptions such as shame and stigma of youth with PSB.

ELIGIBILITY:
Inclusion Criteria:

* Child between the ages of 7-12 who is referred to the treatment program for youth with PSB
* At least one incident of developmentally inappropriate sexual behavior
* Speak and understand English

Exclusion Criteria:

* Court mandate to participate in treatment
* Anticipation of a change of placement within three months
* Have a current diagnosis of a developmental disorder, schizophrenia, bipolar disorder, or intellectual disability

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Attendance in Treatment | 18 weeks
  Completed number of treatment sessions
Provider Rated Engagement | 18 weeks
  Measure completed weekly from the lead therapist regarding each family's participation in the treatment session

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | 18 weeks
  The CSQ-8 is an 8-item reliable and valid outcome measure that assesses for client satisfaction with treatment services. The CSQ-8 has no subscales and reports a single score measuring a single dimension of overall satisfaction with treatment. Higher scores indicate a stronger level of satisfaction.
Working Alliance Inventory (WAI-SR; WAI-CA) | 18 weeks
  Treatment alliance between the therapist and family will be measured using the Working Alliance Inventory - Short Revised (WAI-SR) and Working Alliance Inventory - Children and Adolescents (WAI-CA). The WAI-SR and WAI-CA assesses the therapeutic alliance between a child and their caregiver with the therapeutic provider. This form will be completed by both caregiver and child at 1-month and discharge. Both the WAI-SR and WAI-CA have demonstrated high levels of internal consistency and external validity. Higher scores represent a higher level of treatment alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Shields, PHD, Principal Investigator — University of Oklahoma
Locations (1):
- CCAN Cares Clinic/OU Child Study Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No